CLINICAL TRIAL: NCT00370786
Title: Effect of Intravitreal Bevacizumab on Non -Age-Related Macular Degeneration (AMD) Related Choroidal Neovascularization (CNV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: ophthalmic research center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8543
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2008-07

CONDITIONS: Choroidal Neovascularization
Keywords: Choroidal neovascularization (CNV); Bevacizumab; Non AMD; High myopia; angioid streaks; Ocular histoplasmosis; Idiopathic
MeSH Terms: conditions — Choroidal Neovascularization; Angioid Streaks | interventions — Bevacizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab

SUMMARY:
To evaluate the effect of bevacizumab for treatment of non-AMD choroidal neovascularization (CNV); eg:angioid streaks, ocular histoplasmosis, high myopia, idiopathic,etc

ELIGIBILITY:
Inclusion Criteria:

* Cases with subfoveal or juxtafoveal CNV due to a non-AMD related cause.

Exclusion Criteria:

* Evidence of AMD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-11; Primary Completion 2007-11 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months

SECONDARY OUTCOMES:
central macular thickness | 6 months
leakage in fluorescein angiography | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh, MD, Tehran, Tehran Province, Iran